CLINICAL TRIAL: NCT06115863
Title: Effect of Early Cognitive Stimulation Interventions on Delirium Among Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: prevention of delirium in ICU
Record Dates: First submitted 2023-09-12; First posted 2023-11-03 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Delirium
Keywords: Early cognitive stimulation; critically ill patients
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial with two parallel groups will be used in the current study.
Who Masked: Outcomes Assessor
Masking Description: Single blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo group (Active Comparator): Delirium will be assessed for patients in the control group twice per day for five consecutive days' pre and post conventional nursing care.
  The researcher will observe the conventional nursing care provided by CCNs in the study setting which may affect delirium incidence twice daily for five consecutive days. These traditional nursing practices may include a close conversation between the nurse and the patient, patient re-orientation, such as providing information about time, date, and location, tactile stimulation during various procedures, and changing patients' positions.
  Interventions: Other: Early Cognitive Stimulation Interventions
- early cognitive stimulation Interventions group (Experimental): Beginning on the first day of the patient's admission to the ICU, the early cognitive stimulation interventions will be implemented for nearly 45 minutes twice daily for five days. One session will be conducted during the morning shift and the other during the evening shift. Each session will include the following:
  1. Cognitive stimulation activities will be administered to patients in the intervention group by a member of his family for 15 minutes twice a day for five consecutive days.
  2. Cognitive training exercises: The researcher will carry out these exercises for a total of 300 minutes over the course of five days, splitting the time between 30 minutes in the morning shift and 30 minutes in the evening shift.
  Interventions: Other: Early Cognitive Stimulation Interventions

INTERVENTIONS:
Other: Early Cognitive Stimulation Interventions — early cognitive stimulation interventions refer to multi-dimensions of stimulative evidenced-based interventions, which are done during the first 24 hours from patient admission to the ICU. They are designed to stimulate cognitive function domains that are impacted by delirium such as attention, registration, recall, and language.

SUMMARY:
Delirium is an acute change in attention and awareness that develops over a relatively short time interval and associated with additional cognitive deficits such as memory deficit, disorientation, or perceptual disturbances.

Delirium negative impact has been widely documented in the medical literature. It has been associated with increased mortality and morbidity, longer hospital stays, increase health care costs, and a longer duration of MV.

Delirium in the ICU can be prevented and treated with a combination of pharmaceutical and non-pharmaceutical interventions.

Cognitive interventions, as part of a delirium prevention strategy, are specific therapies focusing on the domains of cognitive functioning impacted by delirium such as orientation, attention, registration, recall and language.

Cognitive stimulation interventions such as orienting patients to the date, time and place, visual and auditory stimulations that focused on specific domains (orientation and registration). In addition, cognitive stimulation included cognitive training and stimulation exercises that focus on specific domains (attention, language, recall, and registration) such as analyzing exercise, recalling exercise, and cognitive-training exercises by using mobile applications .

The involvement of family members in the cognitive stimulation of critically ill patients is an underutilized resource that may benefit patients as well as gain a sense of control and purpose.

DETAILED DESCRIPTION:
Nurses have direct contact with patients 24 hours a day, so they are in an ideal position to prevent, detect, manage, and care for patients who have delirium. The identification of predisposing or precipitating variables must be a part of the nursing intervention in order to reduce the likelihood of delirium occurring. When possible, nurses can help identify at-risk individuals and lower risk. Although a regular nursing assessment and good observational skills combined with a strong therapeutic relationship can enable nurses to recognize sudden changes in attention or consciousness, which are typical indications of delirium.

Although the effects of cognitive stimulation interventions have been extensively studied in the prevention of delirium for ICU patients, there are few studies have implemented to assess its effects when it is applied early within the first 24 hours from ICU admission worldwide, and up to our knowledge there are no national studies that have been conducted to assess early effects of such interventions on delirium in ICU. Therefore, this study will be conducted to evaluate the effect of early cognitive stimulation interventions on delirium in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years.
* Newly admitted patients not more than 24 hours.
* Patient's Richmond Agitation Sedation Scale (RASS) from -1 to +1.

Exclusion Criteria:

* Patient with pre-existing brain injury and cognitive impairment.
* Patient who is delirious on admission positive for Confusion Assessment Method for the ICU 7 (CAM ICU 7).
* Patient with hearing and visual impairment.
* Patients who is Hemodynamically unstable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2025-08-17 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
1. To assess the effect of early cognitive stimulation interventions on delirium among 65 critically ill patients by use CAM -ICU 7. | 5 day from patients' admission to ICU.
  Critically ill patients who undergo early cognitive stimulation interventions have a significantly lower risk of incidence delirium than those who do not. Delirium will be assessed for patients by use the Confusion Assessment Method for the ICU 7 (CAM-ICU 7).
2. To investigate the effect of early cognitive stimulation interventions on delirium severity among 65 critically ill patients. | 5 days from patients' admission to ICU.
  Critically ill patients who undergo early cognitive stimulation interventions show improved the delirium severity scoring compared to those who do not. the measurement tool for delirium severity is CAM-ICU 7

SECONDARY OUTCOMES:
1. To investigate the effect of early cognitive stimulation interventions on patient's length of ICU stay. | immediately after the intervention.
  Critically ill patients who undergo early cognitive stimulation interventions have a significantly shorter length of ICU stay than those who do not.

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Younes Othman Ramadan, ASS-PROF, Study Director — Damanhour University
Locations (1):
- Not Found, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all content of protocol will be accessible to public
Supporting Information: Study Protocol, SAP
Time Frame: just i finish my data entry
Access Criteria: aims , inclusion criteria and methodology

REFERENCES:
- [Background] Hering KG, Mitrovic D. [Diseases of the brachial plexus after surgery and irradiation of breast cancer (author's transl)]. Strahlentherapie. 1981 Feb;157(2):86-90. German. PMID 7222136
- [Background] Deemer K, Myhre B, Oviatt S, Parsons M, Watson M, Zjadewicz K, Soo A, Fiest K, Posadas-Calleja J. Occupational therapist-guided cognitive interventions in critically ill patients: a feasibility randomized controlled trial. Can J Anaesth. 2023 Jan;70(1):139-150. doi: 10.1007/s12630-022-02351-9. Epub 2022 Nov 16. PMID 36385466